CLINICAL TRIAL: NCT03653845
Title: Adrenal Artery Ablation for Primary Aldosteronism：A Randomized, Parallel, Active-controlled Clinical Trial to Evaluate the Efficacy and Safety of Adrenal Artery Ablation（AAA）in the Treatment of Primary Aldosteronism
Brief Title: Adrenal Artery Ablation for Primary Aldosteronism
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhiming Zhu, Director of the Department of Hypertension & Endocrinology, Daping Hospital, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAA-PA
Record Dates: First submitted 2018-06-07; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Primary Aldosteronism; Hypertension
Keywords: Hypertension; Primary Aldosteronism; Ablation; Adrenal Gland
MeSH Terms: conditions — Hyperaldosteronism; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intevention (Experimental): Patients in this group will be treated with endovascular chemical ablation of adrenal glandp by endovascular injection of dehydrated alcohol. Sequenced antihypertensvie drugs with titrated dosage(amlodipine 5-10 mg/d ; terazosin 2-6mg/d) will be prescribed if home blood pressure (HBP) exceeds ≥160/100 mmHg.
  Interventions: Procedure: Endovascular chemical Ablation of Adrenal Gland; Drug: Sequenced antihypertensvie drugs with titrated dosage
- Control (Active Comparator): Patients in this group will be treated only with sequenced antihypertensvie drugs with titrated dosage(amlodipine 5mg/d→plus spironolactone 20 mg/d→plus spironolactone 40 mg/d→plus spironolactone 60 mg/d→→plus amlodipine 10 mg/ d →plus terazosin 2-6mg / d) if home blood pressure (HBP) exceeds ≥160/100 mmHg.
  Interventions: Drug: Sequenced antihypertensvie drugs with titrated dosage

INTERVENTIONS:
Procedure: Endovascular chemical Ablation of Adrenal Gland — Patients in this group will be treated with partial ablation of adrenal gland by endovascular injection of dehydrated alcohol.
  Arms: Intevention
Drug: Sequenced antihypertensvie drugs with titrated dosage — Patients will be treated with different antihypertensive drugs in two groups.

SUMMARY:
Primary aldosteronism (PA) is one of the most common causes of endocrine and resistant hypertension. Current studies have shown that the activation of the renin-angiotensin-aldosterone system (RAAS) and the increased sympathetic nerve activity in the central or local tissue are the key mechanisms of high blood pressure and its organ damages.

The classical method for diagnosis of primary aldosteronism depends on the detection of peripheral venous blood aldosterone level, which is incapable of accurate positioning diagnosis. On the other hand, the current guidelines recommend that surgery and aldosterone receptor inhibitors were the only treatment for primary aldosteronism. However, only about 35% of aldosterone tumors and a small part of unilateral adrenal hyperplasia can be treated by surgery. More than 60% of idiopathic aldosteronism and bilateral adrenal hyperplasia need long-term drug therapy. However, long-term aldosterone inhibitor treatment may also cause hyperkalemia, male breast hyperplasia, female hirsutism and other adverse reactions.

Therefore, the investigators proposed that endovascular chemical partial ablation of the adrenal gland can lower the aldosterone level, reduce the blood pressure and recover the potassium metabolism balance. In order to confirm the above effects, the investigators conduct an open, prospective, positive controlled study in patients with primary aldosteronism patients (including aldosterone, idiopathic aldosteronism and adrenal hyperplasia). The effects on blood pressure, blood electrolytes, adrenal hormones, metabolic indexes, target organ damages were observed to explore the efficacy and safety of the endovascular ablation of the adrenal gland in the treatment of primary aldosteronism.

ELIGIBILITY:
Inclusion Criteria:

* Primary Aldosteronis diagnosed by increased Renin ratio (ARR) and serum aldosterone levels ≥15 ng / dl, and confirmed by saline injection test or captopril inhibition test.
* Idiopathic aldosteronism, bilateral adrenal hyperplasia, and unilateral adrenal hyperplasia with no superior secretion confirmed with adrenal CT and adrenal venous blood (AVS).
* The patients were diagnosed with aldosteronoma or unilateral adrenal hyperplasia but refused to surgical excision.
* Signed informed consent and agreed to participate in this study.

Exclusion Criteria:

* Aldosterone cancer.
* Hyperkalemia.
* Renal failure or the following history of nephropathy: serum creatinine 1.5 times higher than the upper limit; dialysis history; or nephrotic syndrome.
* Secondary hypertension except the primary aldosteronism.
* Adrenergic insufficiency.
* Heart failure with NYHA grade Ⅱ-Ⅳ grade or unstable angina, severe cardiovascular and cerebrovascular stenosis, myocardial infarction, intracranial aneurysm, stroke and other acute cardiovascular events.
* Acute infections, tumors and severe arrhythmias, psychiatric disorders, drugs or alcohol addicts.
* Liver dysfunction or the following history of liver disease: AST or ALT 3 times higher than the upper limit, liver cirrhosis, history of hepatic encephalopathy, esophageal variceal history or portal shunt history.
* Coagulation dysfunction.
* Pregnant women or lactating women.
* Participated in other clinical trials or admitted with other research drugs within 3 months prior to the trial.
* Any surgical or medical condition which can significantly alter the absorption, distribution, metabolism, or excretion of any study drug.
* Allergy or any contraindications for the study drugs, contrast agents and alcohol.
* Refused to sign informed consent

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Change of 24-h average systolic blood pressure measured at baseline and the end of the trial | 24 weeks
  Difference in the change of 24-h average systolic blood pressure compared with the baseline at the end of the study (24 weeks) between the intervention and control group is to be analysed.

SECONDARY OUTCOMES:
Change of blood electrolytes（serum potassium and natrium in mmol/L）measured at baseline and the end of the trial | 24 weeks
  Difference in the change of blood electrolytes（serum potassium and natrium in mmol/L) compared with the baseline at the end of the study (24 weeks) between the intervention and control group is to be analysed.
Change of plasma aldosterone and 24-h urine aldosterone measured at baseline and the end of the trial | 24 weeks
  Difference in the change of plasma aldosterone and 24-h urine aldosterone compared with the baseline at the end of the study (24 weeks) between the intervention and control group is to be analysed.
Change of plasma renin measured at baseline and the end of the trial | 24 weeks
  Difference in the change of plasma renin compared with the baseline at the end of the study (24 weeks) between the intervention and control group is to be analysed.
Change of 24-h average systolic blood pressure measured at the end of the trial compared with the baseline | 24 weeks
  Change of 24-h average systolic blood pressure compared with the baseline at the end of the study (24 weeks) in the intervention group.
Change of anti-hypertensive regimen assessed at baseline and the end of the trial | 24 weeks
  Difference in the change of anti-hypertensive regimen compared with the baseline at the end of the study (24 weeks) between the intervention and control group is to be analysed.
Change of 24-h average diastolic blood pressure, daytime mean systolic blood pressure, daytime mean diastolic blood pressure, and nighttime average systolic and diastolic blood pressure measured at baseline and the end of the trial | 24 weeks
  Difference in the change of 24-h average diastolic blood pressure, daytime mean systolic blood pressure, daytime mean diastolic blood pressure, and nighttime average systolic and diastolic blood pressure compared with the baseline at the end of the study (24 weeks) between the intervention and control group is to be analysed.
Change of home systolic and diastolic pressure measured at baseline and the end of the trial | 24 weeks
  Difference in the change of home systolic and diastolic pressure compared with the baseline at the end of the study (24 weeks) between the intervention and control group is to be analysed.
Change of office systolic and diastolic pressure measured at baseline and the end of the trial | 24 weeks
  Difference in the change of office systolic and diastolic pressure compared with the baseline at the end of the study (24 weeks) between the intervention and control group is to be analysed.
Change of liver enzymes measured at baseline and the end of the trial | 24 weeks
  Difference in the change of liver enzymes (ALT, AST in IU/L) compared with the baseline at the end of the study (24 weeks) between the intervention and control group is to be analysed.
Change of kidney function measured at baseline and the end of the trial | 24 weeks
  Difference in the change of serum creatinine in umol/L compared with the baseline at the end of the study (24 weeks) between the intervention and control group is to be analysed.
Change of fasting blood glucose and lipids profiles measured at baseline and the end of the trial | 24 weeks
  Difference in the change of fasting blood glucose and lipids profiles (TC, HDL-C, LDL-C, TG) in mmol/L compared with the baseline at the end of the study (24 weeks) between the intervention and control group is to be analysed.
Change of sex hormones measured at baseline and the end of the trial | 24 weeks
  Difference in the change of 17-OH, DHEAS, testosterone and estrogen levels compared with the baseline at the end of the study (24 weeks) between the intervention and control group is to be analysed.
Change of 24-h urine microalbumin, microalbumin/creatinine ratio measured at baseline and the end of the trial | 24 weeks
  Difference in the change of 24-h urine microalbumin, microalbumin/creatinine ratio compared with the baseline at the end of the study (24 weeks) between the intervention and control group is to be analysed.
Change of cardiac parameters assessed by echocardiography (IVSd、IVSs、LVPWd, LVPWs, LVEDD, LVEF, LVM) measured at baseline and the end of the trial | 24 weeks
  Difference in the change of cardiac parameters assessed by echocardiography (IVSd、IVSs、LVPWd, LVPWs, LVEDD, in millimetre(mm), and LVEF(%), LVM in gram) compared with the baseline at the end of the study (24 weeks) between the intervention and control group is to be analysed.
Change of carotid intima-media thickness assessed by carotid ultrasound at baseline and the end of the trial | 24 weeks
  Difference in the change of carotid intima-media thickness(CIMT) in millimetre(mm) compared with the baseline at the end of the study (24 weeks) between the intervention and control group is to be analysed.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The third hospital affiliated to the Third Military Medical University, Chongqing, Chongqing Municipality
  - The third hospital affiliated to the Third Military Medical University, Chongqing